CLINICAL TRIAL: NCT01971788
Title: The MATRIX OCT Substudy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: S.M. Misericordia Hospital (Other)
Responsible Party: Principal Investigator, Andrea Picchi, MD, PhD, S.M. Misericordia Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MATRIXOCT2013
Record Dates: First submitted 2013-10-18; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction, Coronary Stent Thrombosis, Antithrombotic Therapy

ARMS (2):
- Prolonged bivalirudin infusion (Experimental): Bivalirudin infusion is prolonged after the end of primary PCI
  Interventions: Device: Optical Coherence Tomography of the infarct related artery
- Intra-procedural bivalirudin infusion (Active Comparator): Bivalirudin infusion is stopped at the end of primary PCI
  Interventions: Device: Optical Coherence Tomography of the infarct related artery

INTERVENTIONS:
Device: Optical Coherence Tomography of the infarct related artery

SUMMARY:
Residual thrombosis of stent struts may occur after the end of primary angioplasty and determine distal embolization and further myocardial damage. Bivalirudin is considered the most appropriate antithrombotic drug in the setting of primary PCI, but an initial increase in stent thrombosis has been reported. In order to overcome this potential adverse event, a prolonged infusion of bivalirudin after the end of PCI has been proposed.

This aim of this study is to test whether the use of long-term bivalirudin infusion, as compared to the intra-procedural only administration, reduces residual thrombosis of stent struts evaluated by optical coherence tomography (OCT) at the end of primary PCI and at 3-5 days follow-up.

A subgroup of patients enrolled in the MATRIX (Minimizing Adverse haemmhorragic events by TRansradial access site and AngioX study) study will be selected showing the following inclusion criteria:

* patients affected by STEMI undergoing primary PCI with stent implantation and randomised to bivalirudin treatment,
* patients who, in addition to the infarct related lesion, show at least one critical stenosis of other coronary vessels suitable for staged-PCI,
* patients whose anatomy is suitable for OCT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the MATRIX (Minimizing Adverse haemmhorragic events by TRansradial access site and AngioX study) study showing the following features:

  1. patients affected by STEMI undergoing primary PCI with stent implantation and randomised to bivalirudin treatment,
  2. patients who, in addition to the infarct related lesion, show at least one critical stenosis of other coronary vessels suitable for staged-PCI,
  3. patients with a coronary anatomy suitable for OCT evaluation.

Exclusion Criteria:

* The same criteria used in MATRIX (Minimizing Adverse haemmhorragic events by TRansradial access site and AngioX study) study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Minimal Flow Area (MinFA) measured at the end of primary PCI and at 4/5-day follow-up | At the end of primary PCI and 4-5 day later

SECONDARY OUTCOMES:
Change in the number of stent cross sections with a thrombotic area > 10% measured at the end of prymary PCI and at 4/5-day follow-up | Athe end of primary PCI and 4/5 days later

CONTACTS AND LOCATIONS:
Locations (1):
- Misericordia Hospital, Grosseto, Italy, Italy